CLINICAL TRIAL: NCT06310486
Title: The Emergency Call on Drowning: A Registry-based Cohort Study of the Characteristics, Predictors, and Outcomes of Fatal and Non-fatal Drowning
Brief Title: The Emergency Call on Drowning
Acronym: DROWN_CALL
Status: Recruiting | Type: Observational
Sponsor: Prehospital Center, Region Zealand (Other)
Responsible Party: Principal Investigator, Niklas Breindahl, Principal Investigator, Prehospital Center, Region Zealand
Other Study IDs: DROWN_CALL
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Drowning; Drowning; Anoxia; Drowning, Near; Drowning; Asphyxia; Drowning and Nonfatal Submersion; Drowning or Immersion of Unknown Intent; Drowning and Submersion, Undetermined Intent; Drowning and Submersion While in Bath-Tub; Drowning and Submersion While in Natural Water; Drowning and Submersion Due to Sailboat Sinking; Drowning and Submersion Due to Fall Off Ship; Drowning and Submersion While in Swimming-Pool
Keywords: Emergency Medical Service (EMS); Drowning; Emergency Medical Dispatch Centre; Emergency Medical Coordination Centre; Dispatch; Emergency Call; Registry; Database; Epidemiology; Danish Drowning Formula; Danish Prehospital Drowning Data; Utstein
MeSH Terms: conditions — Drowning; Hypoxia; Near Drowning; Asphyxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fatal drowning: These patients experienced a drowning incident and died within 30 days after the incident because of their submersion injury.
  Interventions: Other: Drowning-related OHCA; Other: Drowning-related non-OHCA
- Non-fatal drowning: These patients experienced a drowning incident and survived until 30 days after the incident.
  Interventions: Other: Drowning-related OHCA; Other: Drowning-related non-OHCA

INTERVENTIONS:
Other: Drowning-related OHCA — These patients were involved in a drowning incident (submersion or immersion in liquid) and experienced out-of-hospital cardiac arrest (OHCA), defined as being unconscious and not breathing normally at any time in the prehospital setting. Some of these patients may die as a consequence of the submersion injury (fatal drowning), while others may survive (non-fatal drowning).
Other: Drowning-related non-OHCA — These patients were involved in a drowning incident (submersion or immersion in liquid) but did not experience an OHCA. Some of these patients may die as a consequence of the submersion injury (fatal drowning), while others may survive (non-fatal drowning).

SUMMARY:
This study aims to 1) describe patient-, setting-, and dispatcher-related characteristics in drowning-related emergency calls to the Emergency Medical Dispatch Centre (1-1-2 emergency phone) and 2) factors associated with 30-day survival. The investigators will separately analyse drowning-related out-of-hospital cardiac arrest (OHCA) and drowning-related non-OHCA. If feasible, the investigators will qualitatively analyse the calls to identify and describe potential barriers for an optimal handling strategy.

DETAILED DESCRIPTION:
Previous studies have explored emergency priority levels, emergency call categorisations, barriers to assessing an emergency call, and the effects on the outcome. However, this has never been done specifically for drowning patients. Drowning presents a rare and special circumstance that may be particularly complex for laypeople and medical dispatchers for several reasons. Despite this complexity and medical dispatchers' potential to optimize treatment and improve outcomes in drowning incidents, the characteristics of drowning-related emergency calls have never been explored.

This protocol presents a registry-based cohort study of drowning-related emergency medical calls to the EMDC (1-1-2 emergency phone) with 30-day follow-up.

Data from the national Danish Prehospital Drowning Data will be linked with audio files and electronic data from the EMDC database using the patient's unique civil registration numbers.

The investigators will construct two lists of variables: one list for OHCA and one for non-OHCA emergency calls. Data collection from the EMDC database will consist of three phases.

In phase 1, three independent reviewers will listen to 20 emergency calls on drowning (10 OHCA and 10 non-OHCA) to identify relevant variables from the calls (e.g., presence of key symptoms [since an emergency call often does not contain information regarding the absence of symptoms], communication barriers [anything that comes in the way of receiving and understanding information], pre-arrival instructions to callers etc.).

In phase 2, the same reviewers will listen to 20 other emergency calls (10 OHCA and 10 non-OHCA) and use the lists for data collection to determine the data availability and completeness. This may result in modifications to the lists of variables. The investigators will use the results as a basis for reviewer training and calculate inter-rater reliability.

Once the reviewers' performances are satisfying (defined as Fleiss kappa ≥0.8), the investigators will move to phase 3 and collect data for all the drowning calls. Emergency calls will be stratified as OHCA or non-OHCA calls.

ELIGIBILITY:
Inclusion Criteria:

* Patients at all ages registered in the Danish Prehospital Drowning Data are eligible.

Exclusion Criteria:

* Obvious clinical signs of irreversible death (decapitation, decomposition, post-mortem lividity, post-mortem rigidity)
* A valid Do-Not-Attempt-Resuscitation (DNAR) order or other code status orders limiting life-sustaining therapies
* Missing or corrupted audio files
* Missing identification number
* Missing 30-day survival

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All validated drowning cases registered in the Danish Prehospital Drowning Data will be linked with data from the EMDC database according to a data minimisation principle. Patients are included in the Danish Prehospital Drowning Data if they have experienced a drowning incident between 2016 and 2023, defined as experiencing respiratory impairment from submersion or immersion in liquid.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-related characteristics influencing the 30-day survival | 30 days after the drowning incident
  Describe patient-related characteristics in drowning-related emergency calls to the EMDC (1-1-2 emergency phone)
Setting-related characteristics influencing the 30-day survival | 30 days after the drowning incident
  Describe setting-related characteristics in drowning-related emergency calls to the EMDC (1-1-2 emergency phone)
Caller-related characteristics influencing the 30-day survival | 30 days after the drowning incident
  Describe caller-related characteristics in drowning-related emergency calls to the EMDC (1-1-2 emergency phone)
Dispatcher-related characteristics influencing the 30-day survival | 30 days after the drowning incident
  Describe dispatcher-related characteristics in drowning-related emergency calls to the EMDC (1-1-2 emergency phone)

CONTACTS AND LOCATIONS:
Overall Officials: Helle Collatz Christensen, MD, PhD, Ass. Prof., Study Director — Prehospital Center, Region Zealand
Locations (1):
- Prehospital Center Region Zealand, Næstved, Denmark

IPD SHARING:
Plan to Share IPD: No
The datasets used and analysed during the current study are available from the corresponding author upon reasonable request.

REFERENCES:
- [Background] Breindahl N, Wolthers SA, Jensen TW, Holgersen MG, Blomberg SNF, Steinmetz J, Christensen HC; Danish Cardiac Arrest Group. Danish Drowning Formula for identification of out-of-hospital cardiac arrest from drowning. Am J Emerg Med. 2023 Nov;73:55-62. doi: 10.1016/j.ajem.2023.08.024. Epub 2023 Aug 15. PMID 37619443
- [Background] Breindahl N, Wolthers SA, Moller TP, Blomberg SNF, Steinmetz J, Christensen HC; Danish Drowning Validation Group. Characteristics and critical care interventions in drowning patients treated by the Danish Air Ambulance from 2016 to 2021: a nationwide registry-based study with 30-day follow-up. Scand J Trauma Resusc Emerg Med. 2024 Mar 6;32(1):17. doi: 10.1186/s13049-024-01189-y. PMID 38448994